CLINICAL TRIAL: NCT04912505
Title: ASPirin in Immune thRombocytopenia Patients With Cardiovascular disEase
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/19/0509
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Purpura, Thrombocytopenic
Keywords: Immune thrombocytopenia; aspirin; pharmacodynamics; proof-of-concept study
MeSH Terms: conditions — Purpura, Thrombocytopenic; Purpura, Thrombocytopenic, Idiopathic | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Single arm with sequential variations of daily aspirin intake time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Sequential variations of daily aspirin intake time
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Run-in phase during one week with daily aspirin intake at 8 AM; visit 1: blood sampling at H24 and H2; intermediate phase (two weeks): daily aspirin intake at 8 PM; visit 2: blood sampling at H12; then daily intake of aspirin at the time preferred by the patient and study end visit 2 weeks after visit 2

SUMMARY:
The incidence of immune thrombocytopenia increases with older age. This population is at risk for arterial thrombosis. Due to an increased turn-over of platelets, low-dose aspirin once daily may be insufficient in this population to protect against arterial thrombosis. This study is aimed at assessing the pharmacodynamics of aspirin once daily on platelet function in these patients.

DETAILED DESCRIPTION:
The incidence of immune thrombocytopenia increases with older age. About 20% of patients who develop immune thrombocytopenia are exposed to low-dose aspirin for arterial thrombosis prophylaxis. Moreover, immune thrombocytopenia patients have an increased risk for developing arterial thrombosis as compared with matched controls from the general population. Because ITP patients have an increased turn-over of platelets and aspirin is an irreversible inhibitor of cyclooxygenase-1, aspirin taken once daily may be insufficient to provide stable inhibition of platelet function. This has been demonstrated in myeloproliferative neoplasms with a higher platelet turn-over as well; aspirin is given twice daily to these patients. In immune thrombocytopenia, epidemiological findings sustain this assumption because aspirin is not associated to an increased risk of bleeding. The primary aim of this study is to assess the residual platelet function after 75 mg aspirin intake (H24). Secondary objectives are to assess the kinetics of platelet function after daily 75 mg aspirin intake and the relation with arterial thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* non-treated immune thrombocytopenia or immune thrombocytopenia with stable treatment (at least 1 month)
* treated with aspirin daily for a cardiovascular disease; stable platelet count < 100 x 109/L
* at least one month following an arterial thrombosis
* no other antiplatelet drug and anticoagulant
* female patient with childbearing potential must have acceptable method of birth control
* affiliated or benefiting from public health insurance

Exclusion Criteria:

* opposition to participate
* adults under guardianship or other legal protection
* deprived of their liberty by judicial or administrative decision
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Thromboxane B2 | 24 hours
  Platelet production of thromboxane B2 24 hours after a 75 mg aspirin intake

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MOULIS, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No